## **Study Identification**

ClinicalTrials.gov ID: NCT03119025 Unique Protocol ID: IFCI-04/10/2015

Brief Title: Autologous Dendritic Cell Vaccine for Treatment of Patients with

Chronic HCV-Infection

Official Title: Safety/Efficacy of Vaccination with Autologous Dendritic Cells Pulsed with Recombinant HCV-Antigens (Core and NS3) for Treatment of

Patients with Chronic HCV-Infection

The protocol was approved by the Ethics Committee of the Institute of Fundamental and Clinical Immunology (approval number: no 88, 04/10/2015)

**April 10, 2015** 

## Statistical Analysis Plan

Data will be analyzed using Statistica 9.0 software. The results of statistical analysis will be presented as median and interquartile range. The Mann–Whitney test (for independent samples;  $p_U$ ) and Wilcoxon test (for dependent samples;  $p_W$ ) will be applied, and differences with p less than 0.05 will be considered statistically significant. Correlation analysis will be conducted by Spearmen's rank-order correlation ( $R_S$ ).